CLINICAL TRIAL: NCT01722448
Title: Nutritional Prevention of Exertional Muscle Dysfunction
Acronym: MUSREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 12-0504
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Muscle Dysfunction; Exertional Rhabdomyolysis; Muscle Strength
Keywords: muscle; muscle dysfunction; choline; exercise; exertional rhabdomyolysis; rhabdomyolysis
MeSH Terms: conditions — Motor Activity; Rhabdomyolysis | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Choline (Experimental): Phosphatidyl choline
  Interventions: Dietary Supplement: Choline
- Placebo (Placebo Comparator): Vegetable oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Choline — 4 capsules with 480 mg choline per day
  Arms: Choline
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The investigators want to find out whether a choline supplement can protect muscle health in young men with very common genetic vulnerabilities. Men, who respond to a brief, but intense set of arm exercise and have a common genetic profile, will be asked to use a choline supplement for three weeks and a placebo for three weeks. Before the begin of the supplementation study and after 3 and 6 weeks the investigators will test response to the exercise challenge and ask that all consumed foods are recorded.

DETAILED DESCRIPTION:
An initial screening questionnaire will determine general eligibility. The investigators will screen white young males with low to moderate choline intake (<450 mg/d) for CK response to exercise (high/low) by having them do intense eccentric exercise (12 elbow flexor contractions of non-dominant arm with dumbbell at 100% maximal lift capacity) and then 72 hours (3 days) later draw 250 μl capillary blood by finger stick for CK, metabolomic and genetic measurements.

The investigators plan to recruit 30 CK responders with an 1958 A allele of the methylenetetrahydrofolate dehydrogenase 1 (MTHFD1), which is present in about 60% of Caucasian males.

All participants will be asked to complete on three days 24-hour diet interviews with an online automated program provided by the National Cancer Institute. Participants of the intervention study will also have to be complete interviews on the final three days of the two intervention periods The recruited candidates will do an initial exercise challenge with no intervention, then a second challenge after three weeks with the first supplement (randomized choline or placebo), then a third challenge after another three weeks with the complementary second supplement (choline if they had placebo first, placebo if they had choline first).

Samples identified only by code will be stored indefinitely at the UNC Nutrition Research Institute to permit the analysis of additional genetic markers related to muscle health and choline metabolism when the capacity for the analysis of such markers becomes available. Such analyses may be carried out at the University of North Carolina Nutrition Research Institute (UNC NRI) or at external laboratories providing the service for the PI. Samples will be destroyed once no such additional analyses are intended or feasible anymore or if the investigators do not continue this research. Storage of the samples is not optional.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* choline intake less than 450 mg
* exertional muscle dysfunction
* susceptible genetic profile

Exclusion Criteria:

* severe chronic illness
* limited range of arm motion
* required use of prescription medication
* required use of dietary supplements

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2012-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Creatine Kinase (CK) activity | 3 weeks
  CK activity in response to an exertional challenge will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kohlmeier, MD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Nutrition Research Institute, Kannapolis, North Carolina, United States